CLINICAL TRIAL: NCT01727492
Title: Prevention of Noise-induced Damage by Use of Antioxidants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Principal Investigator, Ethisch Comité UZ Antwerpen, Ethics Comittee UZ Antwerpen, University Hospital, Antwerp
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 12/18/172
Record Dates: First submitted 2012-09-28; First posted 2012-11-16 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2013-11

CONDITIONS: Noise-induced Tinnitus; Noise-induced Hearing Loss
Keywords: prevention; noise-induced tinnitus; noise-induced hearing loss; young population
MeSH Terms: conditions — Tinnitus; Hearing Loss, Noise-Induced

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- sugar pill (Placebo Comparator)
- Antioxidantia (Active Comparator): Dosage: 600mg n-acetylcystein and 200mg magnesium intake: 1 hour before leisure noise exposure above 100dB of at least 30 minutes frequency: 4 separate events (2x placebo, 2x antioxidants)
  Interventions: Drug: Antioxidantia

INTERVENTIONS:
Drug: Antioxidantia
  Arms: Antioxidantia

SUMMARY:
The current study is a dubble-blinde placebo-controlled cross-over study verifying the preventive effect of antioxidants on noise-induced hearing loss (NIHL) and noise-induced tinnitus (NIT). The antioxidants comprise of a mixture of magnesium and n-acetylcystein which should be taken 1h before leisure noise above 100dB for at least 30 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-25 years old
* Temporary tinnitus after noise exposure: loudness >5 on a VAS

Exclusion Criteria:

* middle ear problems
* Allergy for magnesium or n-acetylcystein
* Use of hearing protection when going out

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2012-11

PRIMARY OUTCOMES:
Protection against noise-induced tinnitus due to antioxidants
  Antioxidants protect against temporary threshold shift. The most prevalent cause of noise-induced tinnitus is noise-induced hearing loss. Therefore, it is assumed that the preventive intake of antioxidants prior to a loud event, might protect against threshold shift as well as noise-induced tinnitus.
  A 50% decrease of tinnitus loudness scored on a Visual Analogue Scale (VAS) compared to placebo trials is expected.

SECONDARY OUTCOMES:
Change of tinnitus duration
  It is expected that with the intake of antioxidants noise-induced tinnitus is prevented or reduced after loud music exposure. In addition, it is expected that the tinnitus persistence is shortened compared to the placebo arm.

OTHER OUTCOMES:
Decrease of temporary threshold shift in antioxidant trials compared to placebo trials
  A limited number of participants will have audiological testing (audiometry including high frequency audiometry, speech-in-noise testing and otoacoustic emissions) prior to the musical event as well as the morning after noise exposure in order to measure the effects of antioxidants on the hearing thresholds and hearing performance.

CONTACTS AND LOCATIONS:
Locations (1):
- Antwerp University Hospital, Antwerp, Edegem, Belgium

REFERENCES:
- [Derived] Gilles A, Ihtijarevic B, Wouters K, Van de Heyning P. Using prophylactic antioxidants to prevent noise-induced hearing damage in young adults: a protocol for a double-blind, randomized controlled trial. Trials. 2014 Apr 5;15:110. doi: 10.1186/1745-6215-15-110. PMID 24708640